CLINICAL TRIAL: NCT07339254
Title: Experiences With and Attitudes Towards Immune Checkpoint Inhibitors in Patients With Non-Small Cell Lung Cancer (NSCLC) - A Single Center, Survey-Based Study
Brief Title: Experiences w/ & Attitudes Towards Immune Chckpt Inhibitors in NSCLC Patients Single Center Survey Based Study
Status: Not yet recruiting | Type: Observational
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: 2N-25-8; NCI-2025-09218 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); HS-25-00563; 2N-25-8 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2025-12-23; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Lung Non-Small Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational: Patients complete surveys on study.
  Interventions: Other: Non-Interventional Study

INTERVENTIONS:
Other: Non-Interventional Study — Non-interventional study
  Other Names: Non-Interventional Observational Study; Noninterventional (Observational) Study

SUMMARY:
This study evaluates patient satisfaction with receiving intravenous (IV) and/or subcutaneous (SC) immunotherapy and to assess patient preference for IV immunotherapy administration versus SC immunotherapy administration either at the hospital or at home.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess patient satisfaction with receiving IV immune checkpoint inhibitors, reflecting whether the patient thought that the experience was safe, convenient, comfortable and proceeded smoothly.

II. To assess patient preference for IV versus home SC ICI administration.

OUTLINE: This is an observational study.

Patients complete surveys on study.

ELIGIBILITY:
Inclusion Criteria:

* * Age ≥ 18 years.
* * Patients must have histopathologically/cytologically confirmed non-small cell lung cancer, currently receiving Atezolizumab, Cemiplimab, Durvalumab, Nivolumab, Pembrolizumab (i.e. the patient has already received at least one cycle of therapy)
* * Previous chemotherapy/radiotherapy/targeted/immunotherapy is allowed at any prior timepoint.
* * Ability to understand and the willingness to sign a written informed consent or presence of a surrogate decision maker who can give consent.

Exclusion Criteria:

* * Patients is unable to consent for themselves
* * Patient has not yet completed the 1st cycle of ICI-based therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with non-small cell lung cancer, currently receiving Atezolizumab, Cemiplimab, Durvalumab, Nivolumab, or Pembrolizumab.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Strength of patient perception of Intravenous (IV) Immune Checkpoint Inhibitor (ICI) therapy | At Baseline through study completion, up to 1 year.
  Outcome data will be collected using a questionnaire per study protocol. A Likert scale rating system of Strongly Disagree, Disagree, Neutral, Agree, Strongly Agree will be used. Summaries of data will be descriptive and standard statistical methods (median) will be used to present the results. Pearson's chi-square test, the Mantel-Haenszel test (or corresponding exact tests, if resulting expected numbers are small) will be used; the resulting p-value will be used as an indication of strength of an observed association.
Patient interest in home SC ICI administration vs. IV ICI administration at the infusion center | At Baseline through study completion, up to 1 year.
  Outcome data will be collected using a questionnaire per study protocol. Results will be summarized with point estimates and confidence intervals; p-values, when calculated, will be used to indicate the strength of an observed association (not just the magnitude).

SECONDARY OUTCOMES:
Strength of patient perception of Subcutaneous (SC) Immune Checkpoint Inhibitor (ICI) therapy. | At Baseline through study completion, up to 1 year.
  Outcome data will be collected using a questionnaire per study protocol. A Likert scale rating system of Strongly Disagree, Disagree, Neutral, Agree, Strongly Agree will be used. Summaries of data will be descriptive and standard statistical methods (median) will be used to present the results. Pearson's chi-square test, the Mantel-Haenszel test (or corresponding exact tests, if resulting expected numbers are small) will be used; the resulting p-value will be used as an indication of strength of an observed association.
Strength of patient interest in home IV ICI administration vs. SC ICI administration at the infusion center. | At Baseline through study completion, up to 1 year.
  Outcome data will be collected using a questionnaire per study protocol. A Likert scale rating system of Strongly Disagree, Disagree, Neutral, Agree, Strongly Agree will be used. Summaries of data will be descriptive and standard statistical methods (median) will be used to present the results. Pearson's chi-square test, the Mantel-Haenszel test (or corresponding exact tests, if resulting expected numbers are small) will be used; the resulting p-value will be used as an indication of strength of an observed association.
Transportation and social barriers to obtaining Intravenous (IV) Immune Checkpoint Inhibitor (ICI) therapy. | At Baseline through study completion, up to 1 year.
  Outcome data will be collected using a questionnaire consisting of 7 questions. The proportion of participants who select each possible category will be reported. The proportions should add up to 1.0. Results will be summarized in 2-way contingency tables to display any associations between these transportation responses. The Mantel-Haenszel test will be used to estimate the strength of the associations in each contingency table.
Quality of life while on Immune Checkpoint Inhibitor (ICI) therapy | At Baseline through study completion, up to 1 year.
  Patient-Reported Outcomes Measurement Information System (PROMIS-29 v2.1) will be used. This is a standardized, self-report questionnaire with 29 items measuring core health areas like physical function, pain (interference & intensity), anxiety, depression, fatigue, sleep, and social participation, providing T-scores (mean 50, SD 10) for consistent comparison, used to capture patient-reported quality of life.
Duration of ICI therapy | Through study completion, up to 1 year.
  Collected from the medical record and will be calculated using the start and end dates.
Reason for Discontinuation of ICI therapy. | Through study completion, up to 1 year.
  Collected from the medical record.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Hsu, Principal Investigator — University of Southern California
Locations (2):
- United States (2):
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California